CLINICAL TRIAL: NCT06546215
Title: An Open-label, Randomized, Single-dose (0.25mg), Four-period Fully Replicated Bioequivalence Study of Digoxin Tablet Under Fasted and Fed Conditions in Healthy Subjects
Brief Title: Bioequivalence Study of Digoxin Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BTINT024-BE-01
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digoxin test drug (Experimental): digoxin tablet, 0.25mg, single dose
  Interventions: Drug: Digoxin
- digoxin reference drug (Active Comparator): digoxin tablet, 0.25mg, single dose
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — Administer a single-dose (0.25mg) of either the reference or the test formulation of digoxin tablets.

SUMMARY:
The study followed an open-label, randomized, single-dose (0.25mg), four-period full-replicate design encompassing both fasted and fed conditions. Subjects were randomized into two sequences, labeled as group A (TRTR) and group B (RTRT), for the four sessions. By the use of a random table produced by SAS statistical software, the individuals were assigned at random to administer a single-dose (0.25mg) of either the reference or the test formulation of digoxin tablets. During the fasted study phase, participants were randomly administered digoxin tablets after an overnight fast of a minimum of 10 hours, and fasting continued for 4 hours post dose. During the fed trial, subjects consumed a high-fat breakfast 30 minutes before administering digoxin tablets, which consisted of approximately 500 to 600 kcal of fat, 150 kcal of protein, and 250 kcal of carbohydrates, totaling around 800 to 1000 kcal calories. The breakfast must be finished within 30 minutes. Digoxin tablets were administered to each subject in a single dosage with 240 mL of water. Each subject was assigned equitably and at random to one of the two groups. A 14-day washout period was implemented between each period. In the fasted study, blood samples were collected at various time points: predose, 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours after dosing. Similarly, in the fed study, blood samples were collected at predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours after dosing. Following collection, the samples underwent centrifugation at 1700g for 10 minutes at 4℃. The resulting supernatant was then divided into two aliquots and stored at -80℃ until further analysis was conducted. A validated high-performance liquid chromatography with tandem mass spectrometry (HPLC-MS/MS) method was employed to assess the level of digoxin in plasma samples. The PK analysis of the plasma concentration-time curve was performed using a non-compartmental modeling method with Phoenix WinNonlin software version 8.2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese adults aged no less than 18 years
* A body mass index (BMI) falling within the range of 19.0 to 26.0 kg/m2, and a body weight of no less than 45kg for females and 50kg for males respectively.
* All participants signed the informed consent form after receiving thorough information about the study protocol and agreed to adhere to it.

Exclusion Criteria:

* Allergic to digoxin tablets and other digitalis preparations, or allergic to two or more drugs (or foods);
* Subjects cannot follow a uniform diet ;
* Subjects cannot tolerate venipuncture or have a history of dizziness with needles or blood;
* Subjects with medical history of cardiovascular (e.g., ventricular fibrillation, sinus node block), liver, kidney, endocrine, digestive tract, hematological, respiratory, malignant tumor, mental disorder, or any of the above diseases judged by the investigators as clinically significant;
* Subjects underwent major surgical procedures within 6 months before screening or planned to undergo surgery during the study, and those who underwent surgery affecting drug absorption, distribution, metabolism, or excretion (except appendicitis surgery);
* Screening stage of physical examination, vital signs measurement, cardiogram, heart color to exceed, whole chest is slice examination, laboratory examination, blood routine, routine urine and blood biochemistry, blood coagulation function, thyroid function, blood/urine pregnancy (only female subjects), etc.), the researchers determine abnormal have clinical significance;
* Creatinine clearance rate (Ccr) that is beyond the scope of 80 ~ 120 ml/min (including boundary value);
* Clinically significant abnormal results of hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, or human immunodeficiency virus antibody;
* Long-term (within 3 months before screening) excessive consumption (more than 8 cups per day, 1 cup =200mL) of tea, coffee, or caffeinated beverages; Or consuming any food or beverage (e.g., coffee, strong tea, chocolate, etc.) containing caffeine within 48 hours before the first dose of study medication;
* Consuming any beverage or food containing grapefruit or other substances affecting drug absorption, distribution, metabolism, excretion, etc., within 48 hours before the first dose of medication;
* Use of any medication known to interact with digoxin tablets within 4 weeks before screening;
* Patients who used long-acting estrogen or progestin injection or implant within 6 months before the trial; Use of short-acting contraceptives within 30 days before the trial;
* Subjects who had used any prescription drugs, over-the-counter drugs, herbal medicines, or health supplements within 14 days before the first study medication;
* 3 months before the screening of daily smoking more than 5 pieces, and chosen to the whole experiments cannot accept ban smokers;
* Positive alcohol breath test before first medication use or had consumed more than 14 standard units (SD) per week (1 SD containing 14g of alcohol) in the 6 months prior to screening;
* Subjects who were positive in drug screening before the first drug use or had a history of drug abuse within 1 year before the test;
* Pregnant or lactating women, and male (or their partner) or female subjects who plan to become pregnant throughout the trial and within 3 months after the end of the study;
* Female subjects who had unprotected sex within 14 days before screening;
* Subjects who participated in another clinical trial and took drugs within 3 months before the first dose of the study drug;
* Subjects donating blood or blood loss ≥400mL within 3 months before the first dose of study medication, or planning to donate blood or blood components during the study or within 3 months after the end of the study;
* The investigator believes that any circumstances may affect the provision of informed consent or compliance with the trial protocol, or that the participant's participation in the trial may affect the trial results or their safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
plasma concentration in fasted study. | predose, 0.17, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours
  plasma concentration-time curve
plasma concentration in fed study. | predose and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hours
  plasma concentration in fasted study.

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Xu, Doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China